CLINICAL TRIAL: NCT01235390
Title: Effects of California Walnuts on Vascular Function and Immune Health in Postmenopausal Women
Brief Title: Effects of the Consumption of California Walnuts on Cardiovascular Health
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200917609-1
Record Dates: First submitted 2010-10-28; First posted 2010-11-05 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Cardiovascular Health; Immune Function
Keywords: Postmenopausal women; walnuts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5 g of walnuts (Experimental)
  Interventions: Dietary Supplement: Walnuts
- 40 g of walnuts (Experimental)
  Interventions: Dietary Supplement: Walnuts

INTERVENTIONS:
Dietary Supplement: Walnuts — The consumption of assigned walnuts once a day during 4 weeks

SUMMARY:
The purpose of this study is to determine the effects of the 4-week consumption of California walnuts on vascular function and immune health in postmenopausal women of ages 50-70.

Primary outcome measures:

* vascular endothelial function
* platelet reactivity
* indoleamine 2, 3-deoxygenase (IDO)

Secondary outcome measures:

* relationship of walnut intake to lipoprotein, fatty acids and oxylipins

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of morbidity and mortality in the United States. The initiation and progression of atherosclerotic vascular disease is multifactoral in nature, and includes endothelial dysfunction, triggered by chronic inflammation. The consumption of foods rich in flavonoids and other phytochemicals has been inversely associated with cardiovascular disease risk in several epidemiological studies.

Aging is physiologically associated with a variable decline in several features of the immune function. In fact, immunosenescence, or aging of the immune system, is characterized by a reduced ability to fight infection and mount an adequate immune response once a novel infection is introduced. Both the innate and acquired immune systems can be affected with immune specific cells, cell signaling, cytokine production, and cell surface marker expression being all subject to age-related changes. The immune system cells within the digestive tract are an accessible and ideal target to stimulate immunity and diet-based nutritional interventions represent a non-invasive, relatively low-cost, and effective method of stimulating the immune function thus ultimately improving the antibody production in subjects at risk for immunosenescence. This is also based on the significant and dynamic interaction between luminal nutrients and the overall immune function. The study of nutritional influences on the immune system represents an area of growing interest to nutritionists, food scientists and immunologists. In general terms, dietary components have the potential to be an accessible and effective immune stimulant given the antigen presenting capacity of the intestine.

Due to their age and menopausal status, postmenopausal women are at a greater risk population for developing CVD. Males tend to show greater rates of CVD than pre-menopausal women, while women following menopause show an increase in CVD development. This increase in CVD for postmenopausal women is associated with endothelial dysfunction that becomes worse with age.

Recent studies have reported that consumption of walnuts is associated with beneficial effects in prevention of chronic diseases, such as cardiovascular disease (CVD), by favorably altering human serum profiles (i.e. decrease in LDL cholesterol and triglycerides and increase in HDL cholesterol and apolipoprotein A1). It has been shown that the consumption of walnuts, which mainly contain α-linolenic acid (ALA), L-arginine, and polyphenols, can beneficially alter vascular function and reduce inflammatory biomarkers. For example, Dr. Ros and his colleagues demonstrated that the addition of walnuts to a high-fat meal could improve endothelial function. This favorable influence on vasoactivity has been attributed to the antioxidant and anti-inflammatory properties of certain biofactors found in the walnuts.

In this study, we will focus on defining the potential role of California walnuts and its effects on vascular health and immune function. We will determine whether short term (4 week) consumption of California walnuts, particularly rich in ALA, L-arginine and polyphenols will improve endothelial function, platelet reactivity and immune function in an at-risk population of postmenopausal women 55-70 years of age.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 70 years of age
* Lack of menses in the last year and FSH 23-116.3 mlU/mL
* Subject is willing and able to comply with the study protocols.
* Subject is willing to consume California walnuts daily for four weeks.
* BMI 18.5-34.9 kg/m2
* Weight ≥ 110 pounds

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* Self reported use of anticoagulation agents including NSAIDs
* Self reported use of oral cortisone or other immunosuppressive agents,
* Self reported underlying neoplasia or immunological disease,
* Dislike of walnuts
* Food faddists or those taking a non-traditional diet
* Self reported physical activity restricted or reduced due to chronic health conditions
* Self reported diabetes
* Blood pressure ≥ 160/90 mm Hg
* PFA-100 readings 10 % outside of normal reference range (normal reference range for ADP-Collagen: 71-118 sec; Epinephrine-Collagen: 94-193 sec).
* Self reported renal or liver disease
* Self reported heart disease, which includes cardiovascular events and Stroke
* Self reported Cushing's syndrome
* Self reported chronic/routine high intensity exercise
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Abnormal Liver, CBC or Chemistry panels (laboratory values outside the reference range) if determined to be clinically significant by Dr. M. Eric Gershwin.
* Self reported cancer within past 5 years
* Self reported history of psychiatric disorders i.e. schizophrenia or bi-polar or depression treated with antidepressants within the last 1 year.
* Self reported use of MAOI inhibitor within the last 1 year (e.g. phenelzine (Nardil), tranylcypromine (Parnate), etc)
* Self reported malabsorption
* Self reported anxiety medications
* Self reported routine use of prescription drugs or over-the counter medications, which may potentially modulate the outcome of this study; including antibiotics, aspirin and aspirin-containing formulations, COX-2 inhibitors, antihistamines, corticosteroids, hypertensive medications, such as ACE-inhibitors and beta-blockers.
* Asthma (can be worsened by mild to moderate food allergies).
* Indications of substance or alcohol abuse within the last 3 years
* Use of multi-vitamin and mineral other than a general formula of vitamins and minerals that meet the RDA
* Use of herbal or plant-based supplements; omega-3 fatty acids, and fish oils in the past 3-6 months, and unwilling to discontinue use while participating in the study.
* Self reported nut allergies

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 0 and 4 hours, 4 weeks after
  Endothelial function is assessed by using peripheral arterial tonometry (PAT).

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Hackman, Ph. D, Principal Investigator — University of California, Davis
Locations (1):
- Ragle Human Nutrition Research Center, Davis, California, United States